CLINICAL TRIAL: NCT06648629
Title: Acceptance and Commitment Therapy for HIV+ Hazardous Drinkers: A Randomized Clinical Trial
Brief Title: Acceptance and Commitment Therapy for HIV+ Hazardous Drinkers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); University of Rochester (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-207; R01AA030935 (NIH)
Record Dates: First submitted 2024-07-29; First posted 2024-10-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: HIV-1-infection; Alcohol Drinking
Keywords: HIV; Alcohol; ACT; Treatment
MeSH Terms: conditions — Alcohol Drinking | interventions — Acceptance and Commitment Therapy; Ethanol; Methods

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the following two pre-specified treatment groups: Acceptance and Commitment Therapy or Brief Alcohol Intervention.
Who Masked: Outcomes Assessor
Masking Description: The investigators will have a research staff members who are responsible for administering baseline appts (with randomization) and post-treatment study appointments. The outcome assessor will be blind to intervention condition. Interventionists will not collect any outcome data. Study investigators and the Data Safety Monitoring Board (DSMB) members will be presented with interim data (e.g., study completion reports) that are blinded to treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (ACT) (Experimental): Participants randomized to the ACT arm will receive six, weekly, 30-45-minute ACT intervention sessions delivered via telephone.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Brief Alcohol Intervention (BI) (Active Comparator): Participants randomized to BI will receive two 30-60 minute sessions of a brief alcohol intervention delivered via telephone, two 5-10-minute booster calls, and two 5-minute reminder phone calls.
  Interventions: Behavioral: Brief Alcohol Intervention

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — ACT is a trans-diagnostic treatment that targets experiential avoidance as an underlying factor common to mental and behavioral health problems. Mindfulness skills and values-guided behavioral action plans are used to decrease experiential avoidance and impact a broad array of psychological symptoms via improved psychological acceptance.
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy (ACT)
Behavioral: Brief Alcohol Intervention — The Brief Alcohol Intervention (BI) is a standard intervention for reducing alcohol use in PWH. The BI includes the creation of a drinking agreement, self-monitoring via drinking diary cards, discussion of risky moods/situation, and strategies for managing these moods/situations.
  Other Names: BI
  Arms: Brief Alcohol Intervention (BI)

SUMMARY:
Alcohol consumption is a critical factor in HIV treatment that significantly contributes to poor treatment-related outcomes. Randomized clinical trials (RCTs) of alcohol interventions for people with HIV (PWH) have had limited success, perhaps due to an increasingly recognized co-morbitity of co-occurring hazardous alcohol use and other mental health-related problems among PWH. This has necessitated a shift in the literature towards trans-diagnostic approaches that target core psychological processes that underlie multiple mental health-related problems. One trans-diagnostic mechanism that is relevant to alcohol and other substance use is experiential avoidance (EA)- i.e., repeated, and maladaptive, use of substances and/or other behaviors to escape or avoid unwanted thoughts, feelings, and/or urges. Acceptance and commitment therapy (ACT) targets EA and is an empirically supported treatment for multiple psychological and behavioral health-related outcomes; however there have not been any full-scale RCTs of ACT for alcohol use among any population, including PWH. The investigators recently adapted a telephone-delivered ACT intervention originally developed for smoking cessation, into an intervention for PWH who drink at unhealthy levels (NIH/NIAAA; R34AA026246). This six-session, telephone-delivered ACT intervention for alcohol use showed high feasibility and acceptability in a pilot RCT conducted by our team. The overall objective of this application is therefore to determine if ACT can significantly reduce alcohol use and comorbid symptoms of depression, anxiety, and stress among adult PWH who drink at unhealthy levels. The specific aims are: To determine the relative efficacy of ACT, compared to BI, for reducing alcohol use among PWH (Aim 1) and to determine if ACT has an effect on trans-diagnostic processes that in turn affect alcohol use and other psychological and functional outcomes (Aim 2). The investigators will accomplish these aims by: conducting a remote, RCT in which the investigators randomly assign 300 PWH who drink at unhealthy levels to either the ACT intervention the investigators developed (n = 150), or a BI intervention (n = 150) previously shown to reduce alcohol use among PWH. The investigators will assess alcohol-related outcomes-via self-report and a biomarker- at baseline, post-treatment (7 weeks post-baseline), and again 3-, 6-, and 12-months post-randomization. The investigators will also measure EA to determine if it mediates treatment effects for alcohol use and other psychological and functional outcomes, measured at all timepoints.

DETAILED DESCRIPTION:
Alcohol use has a substantial impact on HIV care. Sixty-seven percent of people with HIV (PWH) report using alcohol in the previous year, 27-40% report drinking at unhealthy levels and ~30% meet criteria for alcohol use disorder (AUD). PWH who are unhealthy drinkers, compared to those who abstain or drink relatively less, experience a significant increase in risk for: mortality, lack of viral suppression, less antiretroviral therapy (ART) utilization and sub-optimal adherence to ART. Unhealthy alcohol consumption has been found to affect nearly every stage of the HIV care continuum, making it a critical factor in HIV treatment.

Randomized clinical trials (RCTs) of alcohol interventions for PWH have had limited success, likely due to lack of attention to co-morbid mental health problems. There have been several reviews of this literature, the most recent of which identified 9 non-overlapping behavioral trials developed specifically to target alcohol use and conducted in the U.S. with adult samples of PWH. Only four of these nine trials resulted in significant effects on alcohol-related outcomes and only two trials had effects on alcohol-related outcomes that were significantly different from the control group at 12-month follow-up. One hypothesized reason for this limited success is an increasingly recognized comorbidity of co-occurring unhealthy alcohol use and other mental health-related problems among PWH. Indeed, up to 63% of PWH meet criteria for both a substance use disorder and another psychiatric disorder-necessitating a shift in the literature towards trans-diagnostic approaches that target core psychological processes that underlie multiple mental health and substance-related problems[. One trans-diagnostic mechanism that is particularly relevant to alcohol and other substance use is experiential avoidance (EA)- i.e., repeated, and maladaptive, use of substances and/or other behaviors to escape or avoid unwanted thoughts, feelings, and/or urges.

Acceptance and commitment therapy (ACT) is a promising trans-diagnostic intervention for PWH.

ACT is a trans-diagnostic treatment that targets experiential avoidance as an underlying factor common to mental and behavioral health problems. Mindfulness skills and values-guided behavioral action plans are used to decrease experiential avoidance and impact a broad array of psychological symptoms via improved psychological acceptance. A recent review of 20 meta-analyses, based on 133 studies, found ACT to be efficacious across multiple psychological and behavioral health-related outcomes including: depression, anxiety, chronic pain, stress, and trans-diagnostic combinations of conditions. Additionally, three meta- analyses have found ACT to be efficacious for smoking and other drug use and there is an emerging literature suggesting ACT is a promising approach for alcohol use. There have not, however, been any full- scale RCTs of ACT for alcohol use among any population, including PWH. Given ACT's potential to improve multiple psychological and alcohol-related problems simultaneously, it holds great promise as an intervention for PWH who are unhealthy drinkers. The investigators recently adapted a telephone-delivered ACT intervention originally developed for smoking cessation, into an intervention for PWH who drink at unhealthy levels (NIH/NIAAA; R34AA026246). With a multidisciplinary team, and with two rounds of input from PWH, the investigators developed a six- session, telephone-delivered ACT intervention for alcohol use and subsequently conducted a pilot feasibility/acceptability RCT. The investigators found high acceptability of the adapted ACT intervention, and evidence of feasibility for conducting a full-scale, remote, RCT.

The overall objective of this application is therefore to determine the relative efficacy of ACT, compared to a standard Brief Alcohol Intervention (BI), for reducing alcohol use and comorbid symptoms of depression, anxiety, and stress among adult PWH who are unhealthy drinkers. The application's specific aims are to:

Aim 1: Determine the relative efficacy of ACT, compared to BI, for reducing alcohol use among PWH.

To achieve this aim, the investigators will: conduct a fully remote, relative efficacy RCT. The investigators will randomly assign 300 PWH who are unhealthy drinkers to either the ACT intervention the investigators developed (n = 150), or a BI intervention (n = 150) previously shown to reduce alcohol use among PWH. The investigators will assess alcohol-related outcomes-via self-report and an objective biomarker (phosphatidylethanol) - at baseline, post-treatment (7 weeks post-baseline), and again 3-, 6-, and 12-months post-randomization. The investigators hypothesize that: the two treatments will have significant, and statistically equivalent, effects on alcohol use at post-treatment and 3-months (H1) and, consistent with a sleeper effect for ACT, the ACT condition will have superior alcohol outcomes at 6- and 12-months post- randomization (H2).

Aim 2: Determine if ACT has an effect on trans-diagnostic processes that in turn affect alcohol use and other psychological and functional outcomes. To achieve this aim, the investigators will: measure EA and determine if it mediates treatment effects for alcohol use and other psychological and functional outcomes. The investigators hypothesize that: ACT will have superior outcomes on stress, anxiety, depression, and functional outcomes at all follow-up timepoints (H3) and that EA will be a significant mediator of all treatment effects, including alcohol use (H4).

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV
* Drink at unhealthy levels based on self-reported answers to the AUDIT-C, referencing drinking over the previous 3 months [score of ≥4 (men) or ≥3 (women) will be used to identify eligible participants]
* on HIV treatment and are
* 18 years or older.
* Read at an 8th grade level
* Can provide a physical address
* Able to provide informed consent

Exclusion Criteria:

* Anyone with a score = 12 on the AUDIT-C will be excluded.
* Anyone with a score ≥20 on the PHQ-9, indicative of severe depression, will be excluded.
* Anyone with a score of ≥15 on the GAD-7, indicative of severe anxiety, will be excluded.

Referrals for mental health treatment will be given to all participants who screen out.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Alcohol use - Frequency | Measured at baseline, 8 weeks post-baseline, 3-, 6- , 12-months post-baseline
  The Timeline Followback will be used to estimate the Number of Drinking Days 30 days prior to study visit appointment
Alcohol Use - Quantity | Measured at baseline, 8 weeks post-baseline, 3-, 6- , 12-months post-baseline
  The Timeline Followback will be used to estimate the Number of Drinks per Drinking Day 30 days prior to study visit appointment
Phosphatidylethanol (PEth) | Measured at baseline, 8 weeks post-baseline, 3-, 6- , 12-months post-baseline
  PEth is a metabolite, formed only in the presence of alcohol use and detectable in dried blood spots for approximately 3-4 weeks. The investigators will use both absolute PEth values and a cutoff of 50 mg/ml to indicate recent unhealthy alcohol use. Based on the consideration of both prevalence of underreport in the sample, the investigators will also consider using a compound measure of PEth+ (PEth ≥50ng/ml) and/or self-reported Alcohol Quantity & Frequency via the AUDIT-C+ (≥4, men; ≥3, women) for any unhealthy alcohol use in the last 21 days as an outcome of interest.

SECONDARY OUTCOMES:
Symptoms of Anxiety | Measured at baseline, 8 weeks post-baseline, 3-, 6- , 12-months post-baseline
  Symptom of anxiety will be measured using the Generalized Anxiety Questionnaire (GAD-7). There are 7 items rated on a scale of 0 (not at all) to 3 (nearly every day). The GAD-7 total score ranges from 0 (no anxiety) to 21 (severe anxiety).
Symptoms of Depression | Measured at baseline, 8 weeks post-baseline, 3-, 6- , 12-months post-baseline
  Symptoms of depression will be measured using the Patient Health Questionnaire (PHQ-9). There are 9 items rated on a scale of 0 (not at all) to 3 (nearly every day). The PHQ-9 total score ranges from 0 (no depression) to 27 (severe depression).
Self-reported levels of Stress | Measured at baseline, 8 weeks post-baseline, 3-, 6- , 12-months post-baseline
  Self-reported levels of stress will be measured using the Perceived Stress Scale (PSS). The PSS consists of 10 items rated on a scale from 0 (never) to 4 (very often). The total score ranges from 0 (indicating no stress) to 40 (indicating high levels of stress).
Biological levels of Stress | Measured at baseline, 8 weeks post-baseline, 3-, 6- , 12-months post-baseline
  Biological levels of stress will be measured by assessing levels of cortisol in samples of nails
Symptoms of Experiential Avoidance | Measured at baseline, 8 weeks post-baseline, 3-, 6- , 12-months post-baseline
  Experiential Avoidance will be measured with the Brief Experiential Avoidance Questionnaire (BEAQ). The BEAQ consists of 15 items rated on a scale from 1 (strongly disagree) to 6 (strongly agree). The total score ranges from 15 (indicating low experiential avoidance) to 90 (indicating high experiential avoidance).

OTHER OUTCOMES:
Alcohol-related Problems | Measured at baseline, 8 weeks post-baseline, 3-, 6- , 12-months post-baseline
  Alcohol-related problems will be measured using the Short Inventory of Problems (SIP). The SIP consists of 15 items rated either 0 (no) or 1 (yes). Higher total scores indicate more alcohol-related problems.
Adherence to HIV Medications | Measured at baseline, 8 weeks post-baseline, 3-, 6- , 12-months post-baseline
  Adherence to HIV medications will be measured using the Visual Analogue Scale (VAS). The VAS is a single-item measure where individuals rate their adherence on a scale from 0% (no adherence) to 100% (perfect adherence). The score is represented as a percentage, with higher scores indicating better adherence to HIV medication.
Functional Impairment | Measured at baseline, 8 weeks post-baseline, 3-, 6- , 12-months post-baseline
  Functional impairment will be assessed using the Brief Inventory of Psychosocial Functioning (B-IPF). The B-IPF consists of 7 items rated on a scale from 1 (not at all) to 6 (very much). The total score ranges from 0 (indicating no functional impairment) to 42 (indicating severe functional impairment).

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Per NOT-AA-22-011, this study will submit and share data with NIAAA Data Archive (NIAAADA), a data repository housed within the National Institute of Mental Health (NIMH) Data Archive (NDA). To this end, the study will fulfill all tasks and expectations associated with NIAAA Data Archive (NIAAADA) Data Sharing Plan (DSP)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will share data in accordance with the default NIAAADA data sharing schedule in accordance with the applicable Data Sharing Terms and Conditions of award.

REFERENCES:
- [Derived] Woolf-King SE, Presutti E, McKenna O, Hahn JA, Abar B, Dahne J, Gump BB, Bendinskas KG, Maisto SA. Acceptance and commitment therapy for people with HIV who drink at unhealthy levels: Protocol for the ACCEPT randomized controlled trial. Contemp Clin Trials. 2025 Dec;159:108130. doi: 10.1016/j.cct.2025.108130. Epub 2025 Oct 24. PMID 41326267